CLINICAL TRIAL: NCT01229722
Title: ARemind: A Personalized System to Remind for Adherence
Acronym: ARemind
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dimagi Inc. (Industry)
Collaborators: Boston University (Other); Boston Medical Center (Other); Harvard Medical School (HMS and HSDM) (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Vikram Sheel Kumar, Chief Medical Officer, Dimagi Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2R44MH080655-02 (NIH); R44MH080655 (NIH)
Record Dates: First submitted 2010-10-26; First posted 2010-10-28 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-02

CONDITIONS: Medication Adherence
Keywords: adherence; reminders; text messages; SMS; mHealth
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beeper (Active Comparator): Patients randomized to the control arm (Beeper) will receive the standard of care at each clinic visit. The subjects will bring their HIV medications every 3 weeks (MEMS measure, pill count) and questioned on their adherence to antiretroviral therapy (ART) in the past 7 days. They will not receive any text messages addressing their adherence to ART between each study visit. Their providers will not be receiving any adherence reports but will be asked to assess their adherence at at the start of the trial (Time 1 or T1) and at subsequent clinic visit scheduled according to a frequency defined by standard of care.
  Interventions: Device: Beeper
- Cell Phone (Experimental): Participants will receive a text message reminder via ARemind at scheduled intervals, with varying frequency. They will also be subject to a remote adherence assessment, over text messages, interactive voice response (IVR), or a remote pill count with assistance over the phone from a counselor. Those who demonstrate lower adherence rates may receive a call from a counselor.
  Interventions: Device: ARemind

INTERVENTIONS:
Device: Beeper — Beepers are handheld portable devices which can be attached to a belt. At regular intervals corresponding to the participant's preferred reminder time, they buzz for a few minutes or until the participant presses a button to stop the buzzing.
  Other Names: ALRT Med Reminder Model PC100
  Arms: Beeper
Device: ARemind — ARemind will personalize reminder messages based on adherence levels and facilitate patient phone calls with social workers/adherence counselors when appropriate. It will also consist of a text-messaging or interactive voice response (IVR) or phone-based pill count remote adherence assessment module.
  Arms: Cell Phone

SUMMARY:
The main aim of this phase II proposal is to continue and complete development of a cellular phone-based system that assists patients with their medication adherence. Adherence reports will be developed with feedback from patients and providers. Software for patients to report their four day recall adherence through text messaging or short message service (SMS) or interactive voice response (IVR) will be built. An initial qualitative study will evaluate the adherence reports, 4-day adherence recalls, and inform the development of content for reminder text messages that could be resistant to user fatigue. A redesigned system will be tested through a 3-week longitudinal study of 15 patients with human immunodeficiency virus/acquired immunodeficiency syndrome (HIV/AIDS). An intervention module will have an analytics engine to track adherence levels and personalize delivery of reminder messages. A clinic appointment module will perform patient appointment reminders. The final system with these modules will be tested through a 24-week efficacy study. A total of 115 patients and providers will be involved in the three user studies.

DETAILED DESCRIPTION:
The specific study aims are described below:

1. Organize the Design, Evaluation, and Implementation Teams: The development of ARemind will be guided by design, evaluation and implementation teams. The design team will build the software architecture and execute the software development with inputs from the user studies. The evaluation team will prepare the institutional review board (IRB) submissions, develop the qualitative instruments, and analyze the qualitative and quantitative data. The implementation team will guide clinical and commercial design aspects including input on the remote adherence assessments, the intervention and clinic appointment modules, and the commercialization plan.
2. Run first user study as a qualitative assessment of patient and provider preferences of ARemind: A web-based adherence report for providers will be developed. Software modules to assess adherence over the phone through 4-day SMS or IVR recalls will be created along with a protocol for performing phone-based unannounced pill counts. The interfaces will be tested as a part of in-depth qualitative semi-structured interviews with 15 providers and 15 patients to guide the system design.
3. Study the content preferences through a second user study: A new version of ARemind (version 2.0) will be built based on the feedback from the first user study. It will include the three remote adherence assessment modules. It will be tested longitudinally for 3 weeks on 15 patients with HIV/AIDS. The patients will use Medication Event Monitoring System (MEMS) software, in the form of MEMS caps, and have weekly clinic visits with adherence counselors who will generate a composite adherence score at each visit. MEMS caps are electronic devices attached to a pill bottle which detect and record the time at which the bottles are opened and closed, using this as an estimate for the number of pills taken. These will be compared to the adherence scores from the remote adherence assessment modules. The patients will give qualitative feedback at each visit on the reminder messages to guide the design of content resistant to user fatigue.
4. Explore the feasibility of ARemind through a third user study: An intervention module with an analytics engine will be built. It will personalize reminder messages based on adherence levels and facilitate patient phone calls with social workers/adherence counselors when appropriate. A clinic appointment reminder module will be created and interfaced with the health information exchange of Boston Medical Center (BMC). A new version of ARemind (version 3.0) will contain these new modules and content improved based upon the second study. ARemind 3.0 will be tested through a 24-week longitudinal study of 70 patients. Thirty five patients will be randomized to use cell phones with ARemind 3.0 (intervention) while 35 patients will use beepers (control). Patients will use MEMS caps for composite adherence scores that will be done at each of their 9 adherence visits during the study. Analysis of feasibility, efficacy, user-fatigue and cost-savings from improved adherence to medications and clinic appointments will be performed in this aim.

NOTE: OF THESE THREE USER STUDIES, THE FIRST TWO ARE CONSIDERED FEASIBILITY STUDIES WHILE THE LAST IS A MORE LONGITUDINAL CLINICAL STUDY. THIS REGISTRATION IN CLINICALTRIALS.GOV DEALS WITH THE THIRD USER STUDY, WHICH IS THE LONGEST, INVOLVES THE MOST PARTICIPANTS, AND DEMONSTRATES THE HIGHEST NUMBER OF INTERVENTIONS.

ELIGIBILITY:
Inclusion Criteria:

* Stable ART (no change of ART for 3 months)
* Greater than 18 years of age
* Self-report adherence < 85%

Exclusion Criteria:

* HIV-infected patients not on ART
* Non-English speaking
* Dementia (via mini mental status exam)
* Incarceration
* Legally blind and./or deaf
* User of pillboxes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vikram S Kumar, M.D., Principal Investigator — Dimagi Inc.; Amy Baranoski, M.D., Principal Investigator — Boston Medical Center
Locations (1):
- Center for HIV/AIDS Care and Research, Boston Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients receiving HIV care at Boston Medical Center were eligible to participate if they were 18+ years of age and prescribed an ART regimen for at least 90 days. Participants were recruited between 2011-2012 during their doctor visit and/or via study flyers in the clinic. Eligibility was confirmed in person or via telephone pre-screening.
Groups:
- Beeper: Patients randomized to the control arm (Beeper) will receive the standard of care at each clinic visit. Although the frequency of the study visit is higher than what is observed in standard of care, the subjects will simply asked to bring their HIV medications every 3 weeks (MEMS measure, pill count) and questioned on their adherence to antiretroviral therapy (ART) in the past 7 days. They will not receive any text messages addressing their adherence to ART between each study visit. Their providers will not be receiving any adherence reports but will be asked to assess their adherence at at the start of the trial (Time 1 or T1) and at subsequent clinic visit scheduled according to a frequency defined by standard of care. The decision to restrict the provision of adherence reports to providers and adherence reinforcement messages to intervention group subjects is appropriate, as it is not yet known whether or not the interventions are more effective than the standard of care.
- Cell Phone: Participants will receive a text message reminder at scheduled intervals, with varying frequency. They will also be subject to a remote adherence assessment, over text messages, interactive voice response (IVR), or a remote pill count with assistance over the phone from a counselor. Those who demonstrate lower adherence rates may receive a call from a counselor.
  ARemind: ARemind will personalize reminder messages based on adherence levels and facilitate patient phone calls with social workers/adherence counselors when appropriate. It will also consist of a text-messaging or interactive voice response (IVR) or phone-based pill count remote adherence assessment module.
Period: Overall Study
Arm/Group | Beeper | Cell Phone
Started | 36 | 34
Completed | 36 | 30
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Population: A total of 70 participants were enrolled, but 4 did not complete the study.
Groups:
- Beeper (Control): Patients randomized to the control arm (Beeper) will receive the standard of care at each clinic visit. Although the frequency of the study visit is higher than what is observed in standard of care, the subjects will simply asked to bring their HIV medications every 3 weeks (MEMS measure, pill count) and questioned on their adherence to antiretroviral therapy (ART) in the past 7 days. They will not receive any text messages addressing their adherence to ART between each study visit. Their providers will not be receiving any adherence reports but will be asked to assess their adherence at at the start of the trial (Time 1 or T1) and at subsequent clinic visit scheduled according to a frequency defined by standard of care. The decision to restrict the provision of adherence reports to providers and adherence reinforcement messages to intervention group subjects is appropriate, as it is not yet known whether or not the interventions are more effective than the standard of care.
- Cell Phone (Intervention): Participants will receive a text message reminder at scheduled intervals, with varying frequency. They will also be subject to a remote adherence assessment, over text messages, interactive voice response (IVR), or a remote pill count with assistance over the phone from a counselor. Those who demonstrate lower adherence rates may receive a call from a counselor.
  ARemind: ARemind will personalize reminder messages based on adherence levels and facilitate patient phone calls with social workers/adherence counselors when appropriate. It will also consist of a text-messaging or interactive voice response (IVR) or phone-based pill count remote adherence assessment module.
- Total: Total of all reporting groups
Arm/Group | Beeper (Control) | Cell Phone (Intervention) | Total
Number analyzed (Participants) | 36 | 30 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.11 (10.49) | 46.73 (9.04) | 47.48 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 27 | 17 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 3 | 14
  Not Hispanic or Latino | 25 | 27 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 5 | 12
  Black | 18 | 21 | 39
  Other | 11 | 4 | 15
Education [Count of Participants; unit: Participants]
  High School or Less | 21 | 20 | 41
  More than High School | 15 | 10 | 25
Employment [Count of Participants; unit: Participants]
  Employed | 6 | 9 | 15
  Unemployed | 30 | 21 | 51
Living [Count of Participants; unit: Participants]
  Homeless | 0 | 3 | 3
  Not homeless | 36 | 27 | 63
Relationship [Count of Participants; unit: Participants]
  Married | 2 | 3 | 5
  Not married | 34 | 27 | 61
Country of Birth [Count of Participants; unit: Participants]
  United States | 28 | 22 | 50
  US Territory | 7 | 3 | 10
  Another Country | 1 | 5 | 6
Primary Language [Count of Participants; unit: Participants]
  English | 35 | 28 | 63
  Non-English | 1 | 2 | 3
Baseline CD4 (per mm3) [Median (Full Range); unit: cells/mm^3] | 523.5 [65 to 1643] | 600 [99 to 1292] | 554.5 [65 to 1643]
Baseline Viral Load [Median (Full Range); unit: copies/mL] | 20.0 [20 to 73728] | 23.5 [20 to 62031] | 20.0 [20 to 73728]

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Anti-retroviral Therapy
Description: MEMS pill caps or boxes will be used to monitor adherence. Each participant will place the drug containing the protease inhibitor, or, if no such drug is being taken, the drug with the highest dosing frequency, inside of a MEMS device, which automatically records each time the pillbox was opened. Participants will bring this to the clinic during their regularly scheduled visits, and those daily measurements will be downloaded to a clinic machine.
Time Frame: Assessed at Baseline and 8 timepoints (every 3 weeks) over 24 weeks. T1 (Baseline), T2 (12 weeks), and T3 (24 weeks) reported here.
Population: A total of 66 Boston Medical Center HIV-positive patients participated in this study. All patients in the study had stable ART prior to enrollment.
Measure: Mean (Standard Deviation); unit: proportion adherence
Groups:
- Beeper (Control): Patients randomized to the control arm (Beeper) received the standard of care at each clinic visit. Although the frequency of the study visit is higher than what is observed in standard of care, the subjects were simply asked to bring their HIV medications every 3 weeks (MEMS measure, pill count) and questioned on their adherence to antiretroviral therapy (ART) in the past 7 days. They did not receive any text messages addressing their adherence to ART between each study visit. Their providers did not receive any adherence reports but were asked to assess their adherence at at the start of the trial (Time 1 or T1) and at subsequent clinic visit scheduled according to a frequency defined by standard of care. The decision to restrict the provision of adherence reports to providers and adherence reinforcement messages to intervention group subjects is appropriate, as it is not yet known whether or not the interventions are more effective than the standard of care.
- Cell Phone (Intervention): Participants received a text message reminder at scheduled intervals, with varying frequency. They potentially received a remote adherence assessment, over text messages, interactive voice response (IVR), or a remote pill count with assistance over the phone from a counselor. Those who demonstrate lower adherence rates received a call from a counselor.
  ARemind: ARemind will personalize reminder messages based on adherence levels and facilitate patient phone calls with social workers/adherence counselors when appropriate. It will also consist of a text-messaging or interactive voice response (IVR) or phone-based pill count remote adherence assessment module.
Arm/Group | Beeper (Control) | Cell Phone (Intervention)
Number analyzed (Participants) | 36 | 30
proportion adherence
  T1 | 0.69 (0.28) | 0.73 (0.25)
  T2 | 0.62 (0.27) | .67 (.24)
  T3 | 0.5 (0.3) | .64 (.26)

2. Primary Outcome: Self-Report
Description: Participants were asked to recall what pills they took and what they missed. Adherence was measured by self report as well as Wise Pill and pill count.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of 7-day adherence
Groups:
- Beeper (Control): Patients randomized to the control arm (Beeper) received the standard of care at each clinic visit. The subjects brought their HIV medications every 3 weeks (MEMS measure, pill count) and were questioned on their adherence to antiretroviral therapy (ART) in the past 7 days. They did not receive any text messages addressing their adherence to ART between each study visit. Their providers did not receive any adherence reports, but were asked to assess their adherence at at the start of the trial (Time 1 or T1) and at subsequent clinic visit scheduled according to a frequency defined by standard of care.
  Beeper: Beepers are handheld portable devices which can be attached to a belt. At regular intervals corresponding to the participant's preferred reminder time, they buzz for a few minutes or until the participant presses a button to stop the buzzing.
- Cell Phone (Intervention): Participants received a text message reminder via ARemind at scheduled intervals, with varying frequency. They also potentially received a remote adherence assessment, over text messages, interactive voice response (IVR), or a remote pill count with assistance over the phone from a counselor. Those demonstrated lower adherence rates received a call from a counselor.
  ARemind: ARemind will personalize reminder messages based on adherence levels and facilitate patient phone calls with social workers/adherence counselors when appropriate. It will also consist of a text-messaging or interactive voice response (IVR) or phone-based pill count remote adherence assessment module.
Arm/Group | Beeper (Control) | Cell Phone (Intervention)
Number analyzed (Participants) | 36 | 30
proportion of 7-day adherence
  T1 | .93 (.1) | .95 (.07)
  T2 | .95 (.07) | .95 (.07)
  T3 | .93 (.1) | .95 (.06)

3. Primary Outcome: Pill Count
Description: During the clinic visits ever 3 weeks over the course of the study, participants will be asked to bring all their pill bottles and count the contents of each bottle with assistance from the study coordinator. This count will be compared with the refill history for that patient from the pharmacy in order to get a sense of how many pills they have taken.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of pills taken as scheduled
Groups:
- Beeper (Control): Patients randomized to the control arm (Beeper) received the standard of care at each clinic visit. The subjects brought their HIV medications every 3 weeks (MEMS measure, pill count) and were questioned on their adherence to antiretroviral therapy (ART) in the past 7 days. They did not receive any text messages addressing their adherence to ART between each study visit. Their providers did not receive any adherence reports but were asked to assess their adherence at at the start of the trial (Time 1 or T1) and at subsequent clinic visit scheduled according to a frequency defined by standard of care.
  Beeper: Beepers are handheld portable devices which can be attached to a belt. At regular intervals corresponding to the participant's preferred reminder time, they buzz for a few minutes or until the participant presses a button to stop the buzzing.
- Cell Phone (Intervention): Participants received a text message reminder via ARemind at scheduled intervals, with varying frequency. They also potentially received a remote adherence assessment, over text messages, interactive voice response (IVR), or a remote pill count with assistance over the phone from a counselor. Those who demonstrated lower adherence rates received a call from a counselor.
  ARemind: ARemind will personalize reminder messages based on adherence levels and facilitate patient phone calls with social workers/adherence counselors when appropriate. It will also consist of a text-messaging or interactive voice response (IVR) or phone-based pill count remote adherence assessment module.
Arm/Group | Beeper (Control) | Cell Phone (Intervention)
Number analyzed (Participants) | 36 | 30
proportion of pills taken as scheduled
  T1 | .59 (.34) | .66 (.41)
  T2 | .62 (.22) | .6 (.24)
  T3 | .58 (.24) | .62 (.25)

ADVERSE EVENTS:
Arm/Group | Beeper | Cell Phone
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/30
Other Adverse Events (participants affected / at risk) | 0/36 | 0/30

LIMITATIONS AND CAVEATS:
There were technical challenges interfacing with the wireless pill management device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No